CLINICAL TRIAL: NCT00469716
Title: Infusion of Hypertonic Saline-hetastarch in Cardiac Surgery
Brief Title: Hypertonic Saline-hetastarch in Cardiac Surgery
Acronym: HH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15789
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Postoperative Cardiorespiratory Failure
Keywords: Fluid balance; respiratory function; cardiac function; inflammation; Cardiopulmonary bypass
MeSH Terms: conditions — Respiratory Aspiration; Inflammation | interventions — Saline Solution, Hypertonic; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Hypertonic saline (7.2%) hetastarch (6 %)(200/0.5)

SUMMARY:
Cardiopulmonary bypass(CPB) is associated with increased fluid extravasation and edema formation. A continuous infusion of a mixture of hypertonic saline/hydroxyethyl starch (HSH)during CPB reduced fluid extravasation and total fluid gain during bypass in an animal model. We hypothesize that a continuous infusion of HSH will reduce fluid load and increase hemodynamic and respiratory functions in patients undergoing coronary artery bypass with CPB.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) is associated with fluid overload and edema formation occasionally resulting in vital organ dysfunction affecting heart, respiratory system , gastrointestinal tract and brain. Hyperosmolar/hyperoncotic preparations (HSH/HSD) have been used in cardiac surgery essentially with the aim to mobilize fluid excess and improve postoperative cardiorespiratory function.Most studies dealing with the administration of HSD or HSH during and after CPB, have used protocols recommended for treatment of severe hypovolemia and shock, that is 4 mL/kg as a bolus, given within minutes.In animal experiments we have used HSD or HSH, 1 mL/kg/h to a total dose of 4 mL/kg during CPB. The use of HSH/HSD reduced the total fluid gain about 50 % and resulted in significantly lower content of tissue water in vital organs as heart and lungs. In the actual clinical trial we hypothesize that a continuous infusion of HSH will reduce fluid load and increase hemodynamic and respiratory functions monitored with the PiCCO system in patients undergoing coronary artery bypass with CPB.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective coronary artery bypass graft surgery

Exclusion Criteria:

* Age <18 years or > 75 years
* BMI< 18 or > 30
* Left ventricular ejection fraction < 40%
* Emergency operations
* Additional valvular diseases
* Impaired renal function
* Serum sodium> 145 mmol/l
* Hematocrit< 30%
* Use of clopidogrel the last 5 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Cardiac output, intrathoracic blood volume, extravascular lung water, global enddiastolic volume | 12 hours

SECONDARY OUTCOMES:
Time to extubation, fluid balance, paO2/FiO2- ratio, frequency of atrial fibrillation, cytokines, time to ICU-release and hospital release.

CONTACTS AND LOCATIONS:
Overall Officials: Marit Farstad, MD, PhD, Principal Investigator — Dep. of Anesthesia and Intensive Care, Haukeland University Hospital, 5021 Bergen , Norway
Locations (1):
- Section for thoracic and cardiovascular surgery, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Mehlhorn U, Geissler HJ, Laine GA, Allen SJ. Myocardial fluid balance. Eur J Cardiothorac Surg. 2001 Dec;20(6):1220-30. doi: 10.1016/s1010-7940(01)01031-4. PMID 11717032
- [Background] Kumle B, Boldt J, Suttner SW, Piper SN, Lehmann A, Blome M. Influence of prolonged cardiopulmonary bypass times on splanchnic perfusion and markers of splanchnic organ function. Ann Thorac Surg. 2003 May;75(5):1558-64. doi: 10.1016/s0003-4975(02)04903-2. PMID 12735579 (Retraction: PMID 21847821 Ann Thorac Surg. 2011 Jul;92(1):412)
- [Background] Harris DN, Oatridge A, Dob D, Smith PL, Taylor KM, Bydder GM. Cerebral swelling after normothermic cardiopulmonary bypass. Anesthesiology. 1998 Feb;88(2):340-5. doi: 10.1097/00000542-199802000-00011. PMID 9477053
- [Background] Harris DN, Bailey SM, Smith PL, Taylor KM, Oatridge A, Bydder GM. Brain swelling in first hour after coronary artery bypass surgery. Lancet. 1993 Sep 4;342(8871):586-7. doi: 10.1016/0140-6736(93)91412-f. PMID 8102722
- [Background] McDaniel LB, Nguyen T, Zwischenberger JB, Vertrees R, Uchida T, Kramer GC. Hypertonic saline dextran prime reduces increased intracranial pressure during cardiopulmonary bypass in pigs. Anesth Analg. 1994 Mar;78(3):435-41. doi: 10.1213/00000539-199403000-00003. PMID 8109757
- [Background] Bueno R, Resende AC, Melo R, Neto VA, Stolf NA. Effects of hypertonic saline-dextran solution in cardiac valve surgery with cardiopulmonary bypass. Ann Thorac Surg. 2004 Feb;77(2):604-11; discussion 611. doi: 10.1016/S0003-4975(03)01486-3. PMID 14759446
- [Background] Farstad M, Haugen O, Kvalheim VL, Hammersborg SM, Rynning SE, Mongstad A, Nygreen E, Husby P. Reduced fluid gain during cardiopulmonary bypass in piglets using a continuous infusion of a hyperosmolar/hyperoncotic solution. Acta Anaesthesiol Scand. 2006 Aug;50(7):855-62. doi: 10.1111/j.1399-6576.2006.01064.x. PMID 16879469